CLINICAL TRIAL: NCT00000712
Title: A Multicenter, Double Blind, Comparative Study of Zidovudine Alone Versus Zidovudine and Acyclovir as Treatment for HIV-Infected Patients With CD4+ Counts Less Than 200 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 063; 11037 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Herpesviridae Infections; Drug Evaluation; Drug Therapy, Combination; Herpesvirus 4, Human; Cytomegalovirus Infections; Acyclovir; Acquired Immunodeficiency Syndrome; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Herpesviridae Infections; Epstein-Barr Virus Infections; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Acyclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Acyclovir

SUMMARY:
Original design: The study's purpose is to compare the effects of zidovudine (AZT) alone to the combination of AZT and acyclovir (ACV) to determine if AZT/ACV is associated with a lower death rate and fewer AIDS related opportunistic infections compared to AZT alone, and to investigate the effect of these treatment plans on cytomegalovirus (CMV) and Epstein-Barr virus (EBV) infections. The study evaluates two doses of AZT used alone versus two doses of AZT combined with ACV. Per 12/11/92 amendment: Another antiretroviral agent may be substituted for AZT.

AZT has been shown to increase the life span of patients with AIDS or advanced AIDS related complex and patients being treated for Pneumocystis carinii pneumonia. Drugs that increase the effectiveness of AZT against HIV may also decrease the need for high doses of AZT. This might reduce some of the negative effects of AZT while not reducing the positive effects.

DETAILED DESCRIPTION:
AZT has been shown to increase the life span of patients with AIDS or advanced AIDS related complex and patients being treated for Pneumocystis carinii pneumonia. Drugs that increase the effectiveness of AZT against HIV may also decrease the need for high doses of AZT. This might reduce some of the negative effects of AZT while not reducing the positive effects.

AMENDED: Patients are randomly assigned to one of two treatment regimens. They receive AZT (or other antiretroviral agent) with or without ACV. Treatment Plan 1: AZT along with placebo at the same time. Treatment Plan 2: AZT and ACV. Therapy is for 104 weeks with an optional extension of 24 weeks or until the end of the study whichever comes first. The maximum duration of therapy for any patient will be 128 weeks. Medication is dispensed on a biweekly basis for the first 4 weeks, then every other month for the remainder of the study. Original design: Patients are randomly assigned to one of four treatment plans to receive AZT alone or AZT and ACV. Medications are given every 4 hours (q4h) orally (PO) while awake (WA). A total of 5 doses/day are given. The per dose schedule for the four plans are: Treatment plan 1: AZT plus placebo (an inactive medication) substituting for ACV. Treatment plan 2: AZT and AZT placebo along with an ACV placebo. Treatment plan 3: AZT and ACV. Treatment plan 4: AZT and AZT placebo and ACV.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Methadone maintenance. Therapies available through expanded access or treatment IND programs unless specifically excluded.
* Allowed within 30 days of study entry:
* Systemic steroids only if given for treatment of Pneumocystis carinii pneumonia.
* Recommended:
* PCP prophylaxis.

Patient must have:

* Recovered from first episode of histologically proven Pneumocystis carinii pneumonia (PCP) or microbiologically proven AIDS-defining opportunistic infection as defined in Centers for Disease Control HIV classification group IV.
* C-1.
* Study entry must be within 120 days of AIDS-defining diagnosis.
* Written documentation of positive antibody to HIV by any federally licensed ELISA test kit. This test should be confirmed by another method, for example, Western blot, radioimmunoassay (RIA), HIV culture.
* Patients cannot be transfusion dependent (requiring blood transfusion more than once per month). The last transfusion must be > 2 weeks before entry.
* AMENDED 90-08-27 to include HIV positive patients with CD4+ count < 200 cells/mm3.

Prior Medication:

Allowed:

* Zidovudine (AZT) for < 365 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Symptomatic visceral or progressive Kaposi's sarcoma (KS) (defined by > 10 new lesions in the 30 days prior to entry).
* Other concurrent neoplasms other than basal cell carcinoma of skin (patients who have been in complete remission for 1 year for a malignancy may be enrolled).
* Malabsorption as defined by persistent diarrhea > 6 stools/day for > 4 weeks. Patients whose sole AIDS-defining condition is constitutional disease as defined in CDC's HIV group IV-A or neurologic disease as defined in CDC's HIV group IV-B or AIDS-associated malignancies as defined in CDC's HIV group IV-C.

Concurrent Medication:

Excluded:

* Acyclovir (ACV) prophylaxis or frequent (> once per month) repeated courses of ACV therapy for herpes simplex virus infection.
* Any concomitant medicine unless required.
* Systemic therapy/prophylaxis/maintenance for AIDS-defining opportunistic infection other than prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Acetaminophen for > 72 hours. Cimetidine.
* Flurazepam.
* Indomethacin.
* Ranitidine.
* Probenecid (if receiving AZT).
* Rifampin.
* Rifampin-related drugs.

Patients with the following are excluded:

* Active opportunistic infections.
* Symptomatic visceral or progressive Kaposi's sarcoma (KS) (defined by > 10 new lesions in the 30 days prior to entry).
* Other concurrent neoplasms other than basal cell carcinoma of skin (patients who have been in complete remission for 1 year for a malignancy may be enrolled).
* Malabsorption as defined by persistent diarrhea > 6 stools/day for > 4 weeks.
* Patients whose sole AIDS-defining condition is constitutional disease as defined in CDC's HIV group IV-A or neurologic disease as defined in CDC's HIV group IV-B or AIDS-associated malignancies as defined in CDC's HIV group IV-C.

Prior Medication:

Excluded:

* Zidovudine (AZT) for > 365 days prior to study entry.
* Excluded within 14 days of study entry:
* Systemic acyclovir (ACV) therapy.
* Excluded within 30 days of study entry:
* Antiretroviral therapy (other than AZT per above).
* Immunomodulating agents.
* Biologic response modifiers.

Excluded within 60 days of study entry:

* Ribavirin.

Prior Treatment:

Excluded within 30 days of study entry:

* Cytotoxic chemotherapy or radiation therapy for Kaposi's sarcoma.

Active substance abuse that would impair compliance with study procedure.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1994-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Collier AC, Study Chair; Hirsch M, Study Chair; Corey L, Study Chair
Locations (8):
- United States (8):
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Massachusetts General Hospital ACTG CRS, Worcester, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Collier AC, Schoenfeld DA, Bourland D, Hirsch M, Davis LG, Corey L. Prospective comparative study of acyclovir (ACV) and zidovudine (ZDV) versus ZDV alone in patients with AIDS. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2;125
- [Background] Ioannidis JP, Collier AC, Cooper DA, Corey L, Fiddian AP, Gazzard BG, Griffiths PD, Contopoulos-Ioannidis DG, Lau J, Pavia AT, Saag MS, Spruance SL, Youle MS. Clinical efficacy of high-dose acyclovir in patients with human immunodeficiency virus infection: a meta-analysis of randomized individual patient data. J Infect Dis. 1998 Aug;178(2):349-59. doi: 10.1086/515621. PMID 9697714